CLINICAL TRIAL: NCT01000701
Title: Inflammation and Acute Coronary Syndromes (ACS) - Novel Strategies for Prevention and Clinical Management
Brief Title: Inflammation and Acute Coronary Syndromes
Acronym: SPUM-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University of Bern (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: SPUM-ACS
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Acute Coronary Syndromes
Keywords: Inflammation; ACS; Prevention; Education; Clinical management
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Thrombus, blood cells, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Subproject 1: Optimize prevention after acute coronary syndromes (ACS) by improving caregiver and patient education (http://elips.hug-ge.ch/eng/index_eng2.htm)

Subproject 2: Discover novel genomic biomarkers of ACS in leukocyte subsets by means of analyzing gene expression profiles and function

Subproject 3: Evaluate novel diagnostic and prognostic biomarkers in soluble form in blood/plasma and urine

Subproject 5: Visualize the vulnerable plaque using intravascular ultrasound/optical coherence tomography (IVUS/OCT) and correlate with outcome and biomarkers

Subproject 7: Characterize the effects of inflammation on progenitor/stem cell-mediated repair after ACS by means of analyzing gene expression profiles and function

ELIGIBILITY:
Inclusion Criteria:

* All patients with age ≥ 18 years presenting within 5 days (preferably within 72 hours) after pain onset with the main diagnosis of ACS (acute myocardial infarction: STEMI /NSTEMI and threatened infarction: unstable angina pectoris), who enter the hospital: The patients show symptoms, which are compatible with angina pectoris (chest pain, dyspnoea) and at least one of the following characteristics:

  * persistent ST-segment elevation or depression, T inversion or dynamic ECG changes, new left bundle branch block (LBBB)
  * Evidence of positive troponin by local laboratory reference values with a rise and/or fall in serial troponin levels
  * known coronary artery disease, specified as status after myocardial infarction, CABG, or PCI or newly documented ≥50% stenosis of an epicardial coronary artery during the initial catheterization

Exclusion Criteria:

* Severe physical disability,
* Dementia (inability to comprehend study), OR
* Less than 1 year of life expectancy (for non-cardiac reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with Acute Coronary Syndromes
  3 control groups:
  * patients with stable coronary artery disease
  * healthy controls (blood bank)
  * peripheral artery occlusive disease (CLI/ALI)
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-10; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) in overall population, defined as composite of cardiac death, myocardial infarction or ischemia-driven revascularization | 30 days and 12 months follow-up

SECONDARY OUTCOMES:
SP2/SP3/SP5: temporal change in biomarkers (12 months). | SP2/SP3/SP5: 13 months
Correlation with plaque burden and neointimal thickness assessed by IVUS/OCT imaging in ST segment elevation myocardial infarction (STEMI) subgroup (13 months) | 13 months

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - University Hospital, Geneva, Geneva, Canton of Geneva
  - University Hospital, Bern, Bern
  - University Hospital, Lausanne, Lausanne
  - University Hospital, Zurich, Zurich

REFERENCES:
- [Derived] Kraler S, Liberale L, Tirandi A, Moriero M, Wang Y, Farag M, Carbone F, Bertolotto MB, Pusterla V, Ramoni D, Ministrini S, Puspitasari YM, Bruno F, Raber L, Di Vece D, Templin C, Muller O, Mach F, Crea F, Camici GG, Lapikova-Bryhinska T, Akhmedov A, von Eckardstein A, Gorog DA, Montecucco F, Luscher TF. The junctional protein associated with coronary artery disease predicts adverse cardiovascular events in patients with acute coronary syndromes at high residual risk. Eur Heart J. 2025 Dec 23:ehaf979. doi: 10.1093/eurheartj/ehaf979. Online ahead of print. PMID 41430589
- [Derived] van der Stouwe JG, Godly K, Kraler S, Godly J, Matter CM, Wenzl FA, von Eckardstein A, Raber L, Mach F, Obeid S, Templin C, Luscher TF, Niederseer D; SPUM-ACS investigators. Body temperature, systemic inflammation and risk of adverse events in patients with acute coronary syndromes. Eur J Clin Invest. 2024 Dec;54(12):e14314. doi: 10.1111/eci.14314. Epub 2024 Sep 30. PMID 39350322
- [Derived] Davies A, Wenzl FA, Li XS, Winzap P, Obeid S, Klingenberg R, Mach F, Raber L, Muller O, Matter CM, Laaksonen R, Wang Z, Hazen SL, Luscher TF. Short and medium chain acylcarnitines as markers of outcome in diabetic and non-diabetic subjects with acute coronary syndromes. Int J Cardiol. 2023 Oct 15;389:131261. doi: 10.1016/j.ijcard.2023.131261. Epub 2023 Aug 11. PMID 37574027
- [Derived] Bruno F, Adjibodou B, Obeid S, Kraler SC, Wenzl FA, Akhtar MM, Denegri A, Roffi M, Muller O, von Eckardstein A, Raber L, Templin C, Luscher TF. Occlusion of the infarct-related coronary artery presenting as acute coronary syndrome with and without ST-elevation: impact of inflammation and outcomes in a real-world prospective cohort. Eur Heart J Qual Care Clin Outcomes. 2023 Sep 12;9(6):564-574. doi: 10.1093/ehjqcco/qcad027. PMID 37197909
- [Derived] Gilgien-Denereaz L, Jakob J, Tal K, Gencer B, Carballo D, Raber L, Klingenberg R, Matter CM, Sudano I, Luscher TF, Windecker S, Muller O, Fournier S, Rodondi N, Mach F, Auer R, Nanchen D. Long-term effects of systematic smoking cessation counselling during acute coronary syndrome, a multicentre before-after study. Swiss Med Wkly. 2022 Jul 18;152:w30209. doi: 10.4414/smw.2022.w30209. eCollection 2022 Jul 18. PMID 35964324
- [Derived] Kraler S, Wenzl FA, Georgiopoulos G, Obeid S, Liberale L, von Eckardstein A, Muller O, Mach F, Raber L, Losdat S, Schmiady MO, Stellos K, Stamatelopoulos K, Camici GG, Srdic A, Paneni F, Akhmedov A, Luscher TF. Soluble lectin-like oxidized low-density lipoprotein receptor-1 predicts premature death in acute coronary syndromes. Eur Heart J. 2022 May 14;43(19):1849-1860. doi: 10.1093/eurheartj/ehac143. PMID 35567560
- [Derived] Klingenberg R, Aghlmandi S, Raber L, Akhmedov A, Gencer B, Carballo D, Nanchen D, Bucher HC, Rodondi N, Mach F, Windecker S, Landmesser U, von Eckardstein A, Hamm CW, Luscher TF, Matter CM. Cysteine-Rich Angiogenic Inducer 61 Improves Prognostic Accuracy of GRACE (Global Registry of Acute Coronary Events) 2.0 Risk Score in Patients With Acute Coronary Syndromes. J Am Heart Assoc. 2021 Oct 19;10(20):e020488. doi: 10.1161/JAHA.120.020488. Epub 2021 Oct 8. PMID 34622666
- [Derived] Weichwald S, Candreva A, Burkholz R, Klingenberg R, Raber L, Heg D, Manka R, Gencer B, Mach F, Nanchen D, Rodondi N, Windecker S, Laaksonen R, Hazen SL, von Eckardstein A, Ruschitzka F, Luscher TF, Buhmann JM, Matter CM. Improving 1-year mortality prediction in ACS patients using machine learning. Eur Heart J Acute Cardiovasc Care. 2021 Oct 27;10(8):855-865. doi: 10.1093/ehjacc/zuab030. PMID 34015112
- [Derived] Rossi VA, Denegri A, Candreva A, Klingenberg R, Obeid S, Raber L, Gencer B, Mach F, Nanchen D, Rodondi N, Heg D, Windecker S, Buhmann J, Ruschitzka F, Luscher TF, Matter CM. Prognostic value of inflammatory biomarkers and GRACE score for cardiac death and acute kidney injury after acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2021 May 25;10(4):445-452. doi: 10.1093/ehjacc/zuab003. PMID 33624028
- [Derived] Winzap P, Davies A, Klingenberg R, Obeid S, Roffi M, Mach F, Raber L, Windecker S, Templin C, Nietlispach F, Nanchen D, Gencer B, Muller O, Matter CM, von Eckardstein A, Luscher TF. Diabetes and baseline glucose are associated with inflammation, left ventricular function and short- and long-term outcome in acute coronary syndromes: role of the novel biomarker Cyr 61. Cardiovasc Diabetol. 2019 Oct 31;18(1):142. doi: 10.1186/s12933-019-0946-6. PMID 31672144
- [Derived] Koskinas KC, Zanchin T, Klingenberg R, Gencer B, Temperli F, Baumbach A, Roffi M, Moschovitis A, Muller O, Tuller D, Stortecky S, Mach F, Luscher TF, Matter CM, Pilgrim T, Heg D, Windecker S, Raber L. Incidence, Predictors, and Clinical Impact of Early Prasugrel Cessation in Patients With ST-Elevation Myocardial Infarction. J Am Heart Assoc. 2018 Apr 13;7(8):e008085. doi: 10.1161/JAHA.117.008085. PMID 29654204
- [Derived] Aghlmandi S, Scharer N, Heg D, Raber L, Zwahlen M, Gencer B, Nanchen D, Carballo D, Carballo S, Juni P, von Eckardstein A, Landmesser U, Rodondi N, Mach F, Windecker S, Matter CM, Luscher TF, Klingenberg R. Thrombus aspiration in acute coronary syndromes: prevalence, procedural success, change in serial troponin T levels and clinical outcomes in a contemporary Swiss cohort. Eur Heart J Acute Cardiovasc Care. 2018 Sep;7(6):522-531. doi: 10.1177/2048872617706480. Epub 2017 Apr 20. PMID 28425755
- [Derived] Klingenberg R, Aghlmandi S, Raber L, Gencer B, Nanchen D, Heg D, Carballo S, Rodondi N, Mach F, Windecker S, Juni P, von Eckardstein A, Matter CM, Luscher TF. Improved risk stratification of patients with acute coronary syndromes using a combination of hsTnT, NT-proBNP and hsCRP with the GRACE score. Eur Heart J Acute Cardiovasc Care. 2018 Mar;7(2):129-138. doi: 10.1177/2048872616684678. Epub 2016 Dec 28. PMID 28029055
- [Derived] Raber L, Klingenberg R, Heg D, Kelbaek H, Roffi M, Tuller D, Baumbach A, Zanchin T, Carballo D, Ostojic M, Stefanini GG, Rodondi N, von Birgelen C, Moschovitis A, Engstrom T, Gencer B, Auer R, Meier B, Mach F, Luscher TF, Juni P, Matter CM, Windecker S; COMFORTABLE and SPUM-ACS Trial Investigators. Safety of Prasugrel Loading Doses in Patients Pre-Loaded With Clopidogrel in the Setting of Primary Percutaneous Coronary Intervention: Results of a Nonrandomized Observational Study. JACC Cardiovasc Interv. 2015 Jul;8(8):1064-1074. doi: 10.1016/j.jcin.2015.03.023. PMID 26205445
- [Derived] Reiser H, Klingenberg R, Hof D, Cooksley-Decasper S, Fuchs N, Akhmedov A, Zoller S, Marques-Vidal P, Marti Soler H, Heg D, Landmesser U, Rodondi N, Mach F, Windecker S, Vollenweider P, Matter CM, Luscher TF, von Eckardstein A, Gawinecka J. Circulating FABP4 is a prognostic biomarker in patients with acute coronary syndrome but not in asymptomatic individuals. Arterioscler Thromb Vasc Biol. 2015 Aug;35(8):1872-9. doi: 10.1161/ATVBAHA.115.305365. Epub 2015 Jun 11. PMID 26069234
- [Derived] Klingenberg R, Heg D, Raber L, Carballo D, Nanchen D, Gencer B, Auer R, Jaguszewski M, Stahli BE, Jakob P, Templin C, Stefanini GG, Meier B, Vogt P, Roffi M, Maier W, Landmesser U, Rodondi N, Mach F, Windecker S, Juni P, Luscher TF, Matter CM. Safety profile of prasugrel and clopidogrel in patients with acute coronary syndromes in Switzerland. Heart. 2015 Jun;101(11):854-63. doi: 10.1136/heartjnl-2014-306925. Epub 2015 Mar 20. PMID 25794517
- [Derived] Auer R, Gencer B, Raber L, Klingenberg R, Carballo S, Carballo D, Nanchen D, Cornuz J, Vader JP, Vogt P, Juni P, Matter CM, Windecker S, Luscher TF, Mach F, Rodondi N. Quality of care after acute coronary syndromes in a prospective cohort with reasons for non-prescription of recommended medications. PLoS One. 2014 Mar 27;9(3):e93147. doi: 10.1371/journal.pone.0093147. eCollection 2014. PMID 24676282
- See also: Related Info — http://www.spum-acs.ch